CLINICAL TRIAL: NCT05118542
Title: Effect of Hyperthyroidism and Its Treatment in Graves' Disease to Early Marker of Atherosclerosis: Review on the Pathway of Insulin Resistance, Lipid, Inflammation, and Endothelial Dysfunction to Pulse Wave Velocity and Carotid Intima-Media Thickness
Brief Title: Effect of Hyperthyroidism and Its Treatment in Graves' Disease to Early Marker of Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Wismandari, Assistant Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-06-0752
Record Dates: First submitted 2021-10-06; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Hyperthyroidism; Graves Disease; Atherosclerosis of Artery; Pathophysiology
Keywords: Hyperthyroidism; Graves Disease; Atherosclerosis; Pathophysiology; Insulin Resistance; Lipid Marker; Inflammatory Marker; PWV; cIMT
MeSH Terms: conditions — Hyperthyroidism; Graves Disease; Atherosclerosis; Insulin Resistance | interventions — Propylthiouracil; Methimazole

STUDY DESIGN:
Intervention Model Description: This study was a single blind, randomized clinical trial study, conducted in Cipto Mangunkusumo National Referral Hospital from January 2019 to August 2020. We included all adult patient aged 18-65 years with newly diagnosed Graves' disease or no prior anti-thyroid drugs medication for more than 1 month, who agreed to participate in the study. The exclusion criteria was pregnancy, history of coronary heart disease, known malignancy, current use of immunosuppressive medication, sepsis, thyroid crisis, or having allergic reaction to anti-thyroid drugs and other severe side effect.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The care providers gave two choice of drug doses to the research assistant. The research assistant then give the participant their drugs based on the assignment from the randomisation.
  The investigator and outcome assessor were blinded to the drugs which the participants received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTU Group (Active Comparator): Propylthiouracil (PTU) was given with adjusted dosage according to patient clinical assessment at every visit by their own endocrinologist
  Interventions: Drug: Propylthiouracil
- Methimazole Group (Active Comparator): Methimazole was given with adjusted dosage according to patient clinical assessment at every visit by their own endocrinologist
  Interventions: Drug: Methimazole

INTERVENTIONS:
Drug: Propylthiouracil — PTU were given to participants with adjusted dosage according to patient clinical assessment at every visit by their own endocrinologist.
  Arms: PTU Group
Drug: Methimazole — methimazole were given to participants with adjusted dosage according to patient clinical assessment at every visit by their own endocrinologist.
  Arms: Methimazole Group

SUMMARY:
During July 2019 to August 2020, a single-blind clinical trial was done to 36 patients with Graves' disease. At the beginning of the study, subjects were accommodated into 2 groups, 17 into PTU groups and 19 into methimazole groups. There were 24 subjects who finished the study, 13 from PTU group and 11 from methimazole group. Blood serum was collected for HOMA-IR, LDL-R, NFĸB, sICAM-1, sVCAM-1 and sE-selectin examination. Meanwhile stiffness and thickness of carotid artery was measured using PWV and cIMT.

DETAILED DESCRIPTION:
This study was a single blind, randomized clinical trial study, conducted in Cipto Mangunkusumo National Referral Hospital from January 2019 to August 2020. We included all adult patient aged 18-65 years with newly diagnosed Graves' disease or no prior anti-thyroid drugs medication for more than 1 month, who agreed to participate in the study. The exclusion criteria was pregnancy, history of coronary heart disease, known malignancy, current use of immunosuppressive medication, sepsis, thyroid crisis, or having allergic reaction to anti-thyroid drugs and other severe side effect. Ethical approval was obtained from the Research Ethics Committee of the Faculty of Medicine, Universitas Indonesia with approval number KET-784/UN.2.F1/ETIK/PPM.00.02/2019.

Study participant was observed every month for 3 months. Anti-thyroid drugs (PTU or methimazole) were given according to true simple randomization with adjusted dosage according to patient clinical assessment at every visit by their own endocrinologist. At baseline visit, first and third month follow up, blood serum was collected to analyse HOMA-IR, LDL-R, NFĸB, sICAM-1, sVCAM-1 and sE-selectin, meanwhile PWV and cIMT were measured using radiofrequency ultrasound examination of carotid arteries.

Categorical data was presented in frequency (%), while numerical data was presented using mean (SD) if normally distributed or median (IQR) if not normally distributed. Correlation Pearson test was performed for normal distributed data and Spearman test for not normal distributed data. To analyze the changes in parameter from baseline, first and third month, repeated ANOVA and General Linear Model test was performed. For not normally distributed data, transformation into normally distributed data was performed and the data was presented as geometric mean (CI 95%).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* Newly diagnosed Graves' disease or no prior anti-thyroid drugs medication for more than 1 month
* Agreed to participate in the study

Exclusion Criteria:

* Pregnancy
* History of coronary heart disease
* Known malignancy
* Current use of immunosuppressive medication sepsis, thyroid crisis
* Having allergic reaction to anti-thyroid drugs and other severe side effect

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity | Change from Baseline to 3 month follow-up
  Pulse wave velocity was measured using radio frequency ultrasound in supine position at both left and right carotid artery
carotid intima media thickness | Change from Baseline to 3 month follow-up
  cIMT was measured using radio frequency ultrasound in supine position at both left and right carotid artery

SECONDARY OUTCOMES:
HOMA-IR | Change from Baseline to 3 month follow-up
  HOMA-IR was calculated from patient fasting blood glucose and fasting insulin, which both were obtained through serum of the patient. Fasting blood glucose was measured using ECLIA methods with Abbott reagent, while fasting insulin were measured using ELISA with D&G International Inc. kit
LDL-R | Change from Baseline to 3 month follow-up
  LDL-R was measured from the patient serum using ELISA with D&G International Inc. kit
NFkB | Change from Baseline to 3 month follow-up
  NFkB was measured from the patient serum using ELISA with Cusabio kit
sICAM-1 | Change from Baseline to 3 month follow-up
  sICAM-1 was measured from the patient serum using ELISA with D&G International Inc. kit
sVCAM-1 | Change from Baseline to 3 month follow-up
  sVCAM-1 was measured from the patient serum using ELISA with D&G International Inc. kit
sE-selectin | Change from Baseline to 3 month follow-up
  sE-selectin was measured from the patient serum using ELISA with D&G International Inc. kit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD would be share under specific request to the investigator

REFERENCES:
- [Background] Bano A, Chaker L, Mattace-Raso FUS, van der Lugt A, Ikram MA, Franco OH, Peeters RP, Kavousi M. Thyroid Function and the Risk of Atherosclerotic Cardiovascular Morbidity and Mortality: The Rotterdam Study. Circ Res. 2017 Dec 8;121(12):1392-1400. doi: 10.1161/CIRCRESAHA.117.311603. Epub 2017 Oct 31. PMID 29089349
- [Background] Rizos CV, Elisaf MS, Liberopoulos EN. Effects of thyroid dysfunction on lipid profile. Open Cardiovasc Med J. 2011;5:76-84. doi: 10.2174/1874192401105010076. Epub 2011 Feb 24. PMID 21660244
- [Background] Bilir C, Gokosmanoglu F, Caliskan M, Cinemre H, Akdemir R. Regression of the carotid intima media thickness by propylthiouracil therapy in Graves' hyperthyroidism. Am J Med Sci. 2012 Apr;343(4):273-6. doi: 10.1097/MAJ.0b013e31822a8284. PMID 21825964
- [Background] Inaba M, Henmi Y, Kumeda Y, Ueda M, Nagata M, Emoto M, Ishikawa T, Ishimura E, Nishizawa Y. Increased stiffness in common carotid artery in hyperthyroid Graves' disease patients. Biomed Pharmacother. 2002 Jul;56(5):241-6. doi: 10.1016/s0753-3322(02)00195-6. PMID 12199623
- [Background] Upala S, Wirunsawanya K, Jaruvongvanich V, Sanguankeo A. Effects of statin therapy on arterial stiffness: A systematic review and meta-analysis of randomized controlled trial. Int J Cardiol. 2017 Jan 15;227:338-341. doi: 10.1016/j.ijcard.2016.11.073. Epub 2016 Nov 9. PMID 27839806
- [Derived] Wisnu W, Alwi I, Nafrialdi N, Pemayun TGD, Pantoro NI, Wijaya CN, Tahapary DL, Tarigan TJE, Subekti I. The Effects of Anti-thyroid Drugs on Lipoproteins and Insulin Resistance in Graves' Disease: A Randomized Clinical Trial. J Lipid Atheroscler. 2024 Sep;13(3):358-370. doi: 10.12997/jla.2024.13.3.358. Epub 2024 Jun 12. PMID 39355401